CLINICAL TRIAL: NCT04204044
Title: A Comparative Study of Myo Inositol and Metformin in Improving Biochemical and Clinical Profile of Patients With Polycystic Ovarian Syndrome; a Randomized Clinical Trial
Brief Title: Comparison of Myoinositol and Metformin in PCO
Acronym: PCO
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rashid Latif Medical College (Other)
Responsible Party: Principal Investigator, Lamia yusuf, Associate Professor, Rashid Latif Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB/2019/027
Record Dates: First submitted 2019-10-22; First posted 2019-12-18 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: PCOS
MeSH Terms: interventions — Metformin; Folic Acid; Inositol

STUDY DESIGN:
Intervention Model Description: GROUP A ( Metformin 500 mg TDS), GROUP B( Myoinositol 2000 mg x BD ), GROUP C.(both metformin,& myoinositol)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment will be assigned to each participant using lottery method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP A ( metformin 500 mg TDS) (Experimental): Life style modifications, Weight reduction and folic acid will be prescribed with metformin 500 mg three times a day
  Interventions: Drug: Metformin Hydrochloride
- GROUP B( myoinositol 2000mg x BD ) (Experimental): Life style modifications, Weight reduction and folic acid will be prescribed with myoinositol 2000 mg two times a day
  Interventions: Drug: Myo-inositol
- GROUP C.(both metformin,& myoinositol) (Experimental): Life style modifications, Weight reduction and folic acid will be prescribed with both metformin,& myoinositol three and two times a day respectively
  Interventions: Drug: Metformin Hydrochloride; Drug: Myo-inositol

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin Hydrochloride is used in PCO
  Other Names: Folic acid
  Arms: GROUP A ( metformin 500 mg TDS); GROUP C.(both metformin,& myoinositol)
Drug: Myo-inositol — Myo inositol used in PCO
  Other Names: Folic Acid
  Arms: GROUP B( myoinositol 2000mg x BD ); GROUP C.(both metformin,& myoinositol)

SUMMARY:
Aim of the study is to compare the effect of myoinositol and metformin in the resumption of the spontaneous menstrual cycle in patients diagnosed with PCOS or having oligo/amenorrhea, reduction in weight and BMI, Improvement in the biochemical and clinical profile of patients with the polycystic syndrome.

The secondary outcome measured will be the rate of pregnancy, miscarriage and term pregnancy among these patients inducted in the study.

It will be a Three-arm prospective double-blind study. this clinical trial will be registered in Public registry. this RCT will be based on CONSORT statement. The patient coming to Gynecology OPD will be randomized into 3 groups GROUP A ( metformin 500 mg TDS), GROUP B( myoinositol 2mg x BD ), GROUP C.(both metformin,& myoinositol).each group will take folic acid and will be asked for lifestyle modifications.

DETAILED DESCRIPTION:
PCOS is a common endocrine disorder in women of reproductive age associated with insulin resistance. Metformin and Myo-inositol being insulin sensitizers improve biochemical parameters. it is aimed to compare the effect of myoinositol and metformin in the resumption of the spontaneous menstrual cycle in patients diagnosed with PCOS or having oligo/amenorrhea, reduction in weight and BMI, Improvement in the biochemical and clinical profile of patients with the polycystic syndrome.

Inclusion criteria: will be based on the Rotterdam criteria of diagnosing PCO. Patients presenting with a history of secondary amenorrhea, irregular menstrual cycle, oligomenorrhea, weight gain, hirsutism, and already diagnosed cases of PCO will be included in this group.

Patients with history of Hyperprolactinemia, Cushing's disease, Hypothyroidism/ Hyperthyroidism, Pregnancy and nursing, Established type 1 or type 2 diabetes mellitus, Any history of drug intake e.g. anti-diabetic or estrogen and progesterone, History of treatment for the same complaint taken in the last 3 months, Unable to come for regular follow-ups, Any pathological cause of bleeding e.g. Fibroid, Polyp, Cervical pathology and known allergic to these drugs would be excluded.

ELIGIBILITY:
Inclusion Criteria:

It will be based on the Rotterdam criteria of diagnosing PCO. Patients presenting with a history of secondary amenorrhea, irregular menstrual cycle, oligomenorrhea, weight gain, hirsutism, and already diagnosed cases of PCO will be included in this group.

Exclusion Criteria:

* Hyperprolactinemia
* Cushing's disease
* Hypothyroidism/ Hyperthyroidism
* Pregnancy and nursing
* Established type 1 or type 2 diabetes mellitus
* Any history of drug intake e.g. anti-diabetic or estrogen and progesterone
* History of treatment for the same complaint taken in the last 3 months
* Unable to come for regular follow-ups
* Any pathological cause of bleeding e.g. Fibroid, Polyp, Cervical pathology
* Known allergic to these drugs

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 126 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-25 (Estimated)

PRIMARY OUTCOMES:
Menstrual cycle regulation | Follow up at 3rd and 6th months
  In the resumption of the spontaneous menstrual cycle in patients diagnosed with PCOS or having oligo/amenorrhea.Improvement in the biochemical and clinical profile of patients with the polycystic syndrome
change in weight | Follow up at 3rd and 6th months
  change in weight and BMI. Weight in Kg(s) and height will be measured in meter(s). BMI will be calculated by dividing weight in Kg with height in meter square

SECONDARY OUTCOMES:
Pregnancy / Miscarriage | 1 year
  The secondary outcome measured will be the rate of conception/pregnancy, miscarriage and term pregnancy among these patients inducted in the study.

CONTACTS AND LOCATIONS:
Overall Officials: LAMIA YUSUF, FCPS,MHPE, Principal Investigator — rlmc lahore
Locations (1):
- Rashid Latif Medical College, Lahore, Punjab Province, Pakistan